CLINICAL TRIAL: NCT04351802
Title: CORonavirus (COVID-19) Diagnostic Lung UltraSound Study
Acronym: COR-DLUS
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 282661
Record Dates: First submitted 2020-04-16; First posted 2020-04-17 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: COVID-19
Keywords: COVID-19; Lung Ultrasound
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Lung ultrasound — Focused lung ultrasound examination

SUMMARY:
This observational study is designed to assess whether focused lung ultrasound examination can improve the diagnosis of COVID-19 lung disease and/or make an alternative diagnosis at a patient's initial hospital presentation. For patients with confirmed COVID-19 the study will also assess whether surveillance lung ultrasound examination can predict clinical outcome over the course of their hospital admission.

DETAILED DESCRIPTION:
Study participants will be screened from and recruited on their entry into the suspected COVID-19 admission pathway at Derriford Hospital, Plymouth, UK. In addition to usual clinical care (including physical exam and observations, blood tests, nasopharyngeal swab for viral PCR testing, and chest x-ray as standard), participants will undergo focused lung ultrasound examination.

Participants who are negative for COVID-19 will be followed up to confirm their final discharge diagnoses, and clinical outcome at either 3 months post-enrolment or discharge from hospital.

Participants who are positive for COVID-19 will have regular focused lung ultrasound examination during their hospital admission in addition to usual clinical care until their treatment for COVID-19 is complete. Their discharge diagnoses and clinical outcome at either 3 months post-enrolment or discharge from hospital (whichever is later).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Suspected or confirmed diagnosis of COVID-19
* Able to provide informed consent to study participation

Exclusion Criteria:

* Age less than 18 years
* Inability to provide informed consent at the time of study enrolment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (greater than or equal to 18 years in age) presenting with suspected COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2020-05-11 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Diagnosis of COVID-19 on lung ultrasound | On day of admission to hospital
  Primary and blinded scorer diagnosis of COVID-19 on lung ultrasound
Difference in diagnosis of COVID-19 on lung ultrasound vs. chest x-ray | On day of admission to hospital
  Primary and blinded scorer diagnosis of COVID-19 on lung ultrasound vs. radiologist-reported chest x-ray findings

SECONDARY OUTCOMES:
Diagnosis of alternative condition to COVID-19 on lung ultrasound vs. chest x-ray | On day of admission to hospital
  Primary and blinded scorer diagnosis of alternative condition on lung ultrasound
Ability of surveillance lung ultrasound to predict clinical trajectory / outcome in patients with COVID-19 | During hospital admission
  Comparison of lung ultrasound findings with clinical markers of COVID-19 disease severity e.g. supplementary oxygen requirements
Consistency of lung ultrasound interpretation in patients presenting with suspected COVID-19 | On day of admission to hospital
  Comparison of primary and blinded scorer evaluation of lung ultrasound scans for consistency of interpretation and diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: John P Corcoran, BMBCh MRCP, Principal Investigator — University Hospitals Plymouth NHS Trust
Locations (1):
- Derriford Hospital, Plymouth, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No